CLINICAL TRIAL: NCT00001017
Title: Comparison of Fluconazole (UK-49,858) and Amphotericin B for Maintenance Treatment of Cryptococcal Meningitis in Patients With Acquired Immunodeficiency Syndrome
Brief Title: Comparison of Fluconazole and Amphotericin B in the Treatment of Brain Infections in Patients With AIDS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Model: Parallel | Purpose: Treatment
Other Study IDs: ACTG 026; 056-158; FDA 12E
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2011-03-14 (Estimated); Status verified 2002-09

CONDITIONS: Meningitis, Cryptococcal; HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Meningitis; Injections, Intravenous; Cryptococcosis; Fluconazole; Administration, Oral; Acquired Immunodeficiency Syndrome; Amphotericin B
MeSH Terms: conditions — Meningitis, Cryptococcal; HIV Infections; AIDS-Related Opportunistic Infections; Meningitis; Cryptococcosis; Acquired Immunodeficiency Syndrome | interventions — Fluconazole; Amphotericin B

INTERVENTIONS:
Drug: Fluconazole
Drug: Amphotericin B

SUMMARY:
To compare the safety and effectiveness of a new drug, fluconazole, with that of the usual therapy, amphotericin B, in the prevention of a relapse of cryptococcal meningitis (CM) in patients with AIDS who have been successfully treated for acute CM in the last 6 months.

Cryptococcal meningitis is a life-threatening infectious complication of AIDS. Because relapse after treatment occurs in over 50 percent of cases, chronic maintenance therapy with intravenous (IV) amphotericin B is usually given. However, amphotericin B is not always effective, has toxic effects, and must be given by the intravenous route. Fluconazole is an antifungal agent that can be given orally and has been shown to be effective against cryptococcal infections in animals and against acute CM in a few AIDS patients. Also, the side effects experienced by over 2000 patients or volunteers given fluconazole have seldom been severe enough to require withdrawal of the drug.

DETAILED DESCRIPTION:
Cryptococcal meningitis is a life-threatening infectious complication of AIDS. Because relapse after treatment occurs in over 50 percent of cases, chronic maintenance therapy with intravenous (IV) amphotericin B is usually given. However, amphotericin B is not always effective, has toxic effects, and must be given by the intravenous route. Fluconazole is an antifungal agent that can be given orally and has been shown to be effective against cryptococcal infections in animals and against acute CM in a few AIDS patients. Also, the side effects experienced by over 2000 patients or volunteers given fluconazole have seldom been severe enough to require withdrawal of the drug.

Patients accepted in the trial are randomly assigned to fluconazole or amphotericin B. Fluconazole is given orally once a day and amphotericin B is given intravenously once a week. Dosages depend on body weight. Medications may be given with amphotericin B to prevent or reduce discomfort from associated side effects. Patients are treated for 12 months and may continue to receive antiviral therapy, radiation therapy for mucocutaneous Kaposi's sarcoma, or preventive therapy for Pneumocystis carinii pneumonia (PCP) during the study.

ELIGIBILITY:
Inclusion Criteria

* HIV infection documented by antibody (ELISA on two occasions or ELISA with Western blot confirmation), p24 antigen testing, or recovery of HIV in culture.

Prior Medication:

Required:

* Minimum total dose of 15 mg/kg of amphotericin B (either alone or in combination with flucytosine) during primary therapy. End of primary therapy within 6 weeks of start of maintenance therapy.
* Allowed:
* Past or present antiviral therapy and prophylaxis for Pneumocystis carinii pneumonia (PCP).
* Pfizer must be notified if the patient is receiving ganciclovir at entry. Allowed with amphotericin B to treat or prevent side effects.
* Antipyretics.
* Hydrocortisone.
* Meperidine.

Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* Clinical evidence of acute or chronic meningitis other than cryptococcosis.
* Allergy or intolerance of imidazoles, azoles, or amphotericin B. Unable to take oral medications reliably.

Patients with the following are excluded:

* Clinical evidence of acute or chronic meningitis other than cryptococcosis.
* Allergy or intolerance of imidazoles, azoles, or amphotericin B.

Prior Medication:

Excluded for more than 7 days after initiation of primary therapy for cryptococcosis:

* Ketoconazole.
* Fluconazole.
* Itraconazole.
* Miconazole.
* Any other systemic imidazole or azole.
* Excluded:
* Intrathecal amphotericin B.
* Coumadin-type anticoagulants.
* Oral hypoglycemics.
* Barbiturates.
* Phenytoin.
* Immunostimulants.
* Investigational drug or approved (licensed) drugs for investigational indications.

Prior Treatment:

Excluded:

* Lymphocyte replacement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330
Dates: Primary Completion 1991-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Armstrong D, Study Chair; Dismukes W, Study Chair; Powderly W, Study Chair
Locations (28):
- United States (28):
  - UCLA CARE Ctr, Los Angeles, California
  - Univ of Miami School of Medicine, Miami, Florida
  - Indiana Univ Hosp, Indianapolis, Indiana
  - Louisiana State Univ School of Medicine, New Orleans, Louisiana
  - Tulane Univ School of Medicine, New Orleans, Louisiana
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Harvard (Massachusetts Gen Hosp), Boston, Massachusetts
  - Beth Israel Deaconess - West Campus, Boston, Massachusetts
  - SUNY / Erie County Med Ctr at Buffalo, Buffalo, New York
  - City Hosp Ctr at Elmhurst / Mount Sinai Hosp, Elmhurst, New York
  - Beth Israel Med Ctr / Peter Krueger Clinic, New York, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Cornell Univ Med Ctr, New York, New York
  - Mem Sloan - Kettering Cancer Ctr, New York, New York
  - Saint Luke's - Roosevelt Hosp Ctr, New York, New York
  - Mount Sinai Med Ctr, New York, New York
  - Univ of Rochester Medical Center, Rochester, New York
  - SUNY - Stony Brook, Stony Brook, New York
  - Jack Weiler Hosp / Bronx Municipal Hosp, The Bronx, New York
  - Montefiore Med Ctr / Bronx Municipal Hosp, The Bronx, New York
  - North Central Bronx Hosp / Bronx Municipal Hosp, The Bronx, New York
  - Bronx Veterans Administration / Mount Sinai Hosp, The Bronx, New York
  - Univ of North Carolina, Chapel Hill, North Carolina
  - Duke Univ Med Ctr, Durham, North Carolina
  - Holmes Hosp / Univ of Cincinnati Med Ctr, Cincinnati, Ohio
  - Univ Hosp of Cleveland / Case Western Reserve Univ, Cleveland, Ohio
  - Ohio State Univ Hosp Clinic, Columbus, Ohio
  - Julio Arroyo, West Columbia, South Carolina

REFERENCES:
- [Background] Saag MS, Powderly WG, Cloud GA, Robinson P, Grieco MH, Sharkey PK, Thompson SE, Sugar AM, Tuazon CU, Fisher JF, et al. Comparison of amphotericin B with fluconazole in the treatment of acute AIDS-associated cryptococcal meningitis. The NIAID Mycoses Study Group and the AIDS Clinical Trials Group. N Engl J Med. 1992 Jan 9;326(2):83-9. doi: 10.1056/NEJM199201093260202. PMID 1727236
- [Background] Powderly WG, Saag MS, Cloud GA, Robinson P, Meyer RD, Jacobson JM, Graybill JR, Sugar AM, McAuliffe VJ, Follansbee SE, et al. A controlled trial of fluconazole or amphotericin B to prevent relapse of cryptococcal meningitis in patients with the acquired immunodeficiency syndrome. The NIAID AIDS Clinical Trials Group and Mycoses Study Group. N Engl J Med. 1992 Mar 19;326(12):793-8. doi: 10.1056/NEJM199203193261203. PMID 1538722
- [Background] Powderly WG, Cloud GA, Dismukes WE, Saag MS. Measurement of cryptococcal antigen in serum and cerebrospinal fluid: value in the management of AIDS-associated cryptococcal meningitis. Clin Infect Dis. 1994 May;18(5):789-92. doi: 10.1093/clinids/18.5.789. PMID 8075272
- [Background] McKinney RE Jr, Maha MA, Connor EM, Feinberg J, Scott GB, Wulfsohn M, McIntosh K, Borkowsky W, Modlin JF, Weintrub P, et al. A multicenter trial of oral zidovudine in children with advanced human immunodeficiency virus disease. The Protocol 043 Study Group. N Engl J Med. 1991 Apr 11;324(15):1018-25. doi: 10.1056/NEJM199104113241503. PMID 1672443